CLINICAL TRIAL: NCT01507701
Title: Pilot Study for the NorCAPITAL Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Vegard Bruun Wyller, Associate Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NorCAPITALps
Record Dates: First submitted 2011-12-22; First posted 2012-01-11 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Fatigue Syndrome
Keywords: adolescents
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clonidine (Experimental)
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Clonidine — 50 micrograms twice a day for 14 days; thereafter 25 microgram clonidine twice a day for 7 days; thereafter discontinuation.

SUMMARY:
The aim of this pilot study for the NorCAPITAL trial is to investigate the feasibility and safety of the drug clonidine in adolescent chronic fatigue syndrome (CFS). Specifically, the investigators wanted to assess appropriate dosage in relation to a) plasma concentration levels of clonidine, b) orthostatic cardiovascular responses (the pulse and blood pressure responses when rising up), and c) reports of possible adverse effects.

A possible beneficial effect of clonidine in adolescent CFS will be investigated in NorCAPITAL, which is a randomized, placebo-controlled, double blind trial.

ELIGIBILITY:
Inclusion Criteria:

* Persisting or constantly relapsing fatigue lasting 3 months or more
* Functional disability resulting from fatigue to a degree that prevent normal school attendance
* Age between 12 and 19 years

Exclusion Criteria:

* Another disease process or current demanding life event that might explain the fatigue
* Another chronic disease
* Permanent use of drugs
* Permanently bed-ridden
* Positive pregnancy test
* Supine systolic blood pressure (SBP) < 85 mm Hg
* Fall in SPB upon standing > 30 mm Hg
* Supine HR < 50 beats/min
* Abnormal ECG

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration level (Cmax and Co) of clonidine | After 14 days of treatment

SECONDARY OUTCOMES:
Orthostatic cardiovascular responses (head-up tilt test) | After 14 days of treatment
Reports of adverse effects | Participants will be followed for the duration of treatment period, an expected average of 14 days
Plasma concentration (Cmax) of clonidine | First day of treatment, approximately 5 hours after the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Bruun Wyller, MD, PhD, Principal Investigator — Oslo University Hospital Rikshospitalet, Dept. of Pediatrics
Locations (1):
- Oslo University Hospital Rikshospitalet, Dept. of Pediatrics, Oslo, Norway

REFERENCES:
- [Derived] Fagermoen E, Sulheim D, Winger A, Andersen AM, Vethe NT, Saul JP, Thaulow E, Wyller VB. Clonidine in the treatment of adolescent chronic fatigue syndrome: a pilot study for the NorCAPITAL trial. BMC Res Notes. 2012 Aug 7;5:418. doi: 10.1186/1756-0500-5-418. PMID 22871021